CLINICAL TRIAL: NCT02188186
Title: Therapeutic Efficacy of Triple Combination of Metformin, DPP4 Inhibitor and Thiazolidinedione in Drug-naïve Korean Type 2 Diabetic Patients
Brief Title: Therapeutic Efficacy of Triple Combination in Drug-naïve Korean Type 2 Diabetic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Triple
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes
Keywords: triple combination; metformin; sitagliptin; thiazolidinedione
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Initial dual combination therapy with sulfonylurea and metfomin. Dose of sulfonylurea (glimepride 2-8 mg) and metfomin (500-2550 mg) can be ecalated at investigator's discreition at every visit.
  Insulin therpy can be added as a rescue therapy at investigator's discreition.
  Interventions: Drug: Conventional treatment
- Initial triple combination treatment (Experimental): Initial dual combination therapy with metformin, sitagliptin (Januvia 100 mg), and lobeglitazone (Duvie 0.5 mg).
  Insulin therpy can be added as a rescue therapy at investigator's discreition.
  Interventions: Drug: Initial triple combination

INTERVENTIONS:
Drug: Initial triple combination — Initial triple combination arm
  Other Names: metformin+sitagliptin (Januvia)+lobeglitazone (Duvie)
  Arms: Initial triple combination treatment
Drug: Conventional treatment — Conventioanl treament with dose escalation
  Other Names: metformin+sulfonylurea with dose escalation
  Arms: Conventional treatment

SUMMARY:
Triple combination of metformin, DPP4 inhibitor and Thiazolidinedione would be a good option in the treatment of drug-naïve Korean type 2 diabetic patients.

DETAILED DESCRIPTION:
Thiazolidionedione, a PPARgamman agonist, is an strong insulin sensitizer. It has shown that durable glucose lowering effect and beta cell preservation. It is an important treatment option in patients with type 2 diabetes.

It has been well established that inhibition of dipeptidyl peptidase-4 (DPP-4) reduces blood glucose levels in both fasting and postprandial states, and preserves pancreatic β-cell function in patients with type 2 diabetes. The mechanism of action of DPP-4 inhibitors is to increase levels of active incretin, glucagon-like peptide-1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP), which stimulate insulin secretion as well as insulin biosynthesis while inhibiting glucagon release from pancreatic islets.

DPP4 inhibitors also have better safety and tolerability profiles (e.g., weight neutrality and less hypoglycemia) compared to other hypoglycemic agents. When considering combination therapy with DPP-4 inhibitors, metformin is the most commonly used agent which has been shown to be effective and well tolerated from previous studies. Besides the glucose lowering effect by reducing hepatic glucose output and improving insulin resistance, metformin without inhibiting DPP-4 activity,also increases active GLP-1 concentrations by 1.5- to 2-fold following an oral glucose load in obese, nondiabetic subjects. Accordingly, this effect of metformin may provide a unique benefit when combined with DPP-4 inhibitors through a substantial enhancement of the incretin axis, which provides effective and potentially additive glycemic improvement.

Because of its favorable pharmacological properties, combination of a DPP-4 inhibitor, metformin, and thiazolidinedione has been increasingly used to achieve rapid glycemic goal with low risk of hypoglycemia and no weight gain, and to delay the need for subsequent regimen changes. DPP-4 inhibitors block DPP-4 enzyme and preserve endogenous incretins whereas metformin increases the active form of GLP-1, both of which may enhance the secretory function of pancreas. However, the response to DPP-4 inhibitors and metformin combination therapy may be different in individuals according to their pancreatic function and insulin resistance status. In fact, previous studies with DPP-4 inhibitors showed different potency in glycemic controls depending on various patient characteristics including severity of diabetes and the use of other antidiabetic drug.Consequently, it would be clinically important to investigate effect of this triple combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 9-12%
* No treatment with insulin or oral agents for recent 6 months
* 20 ≤ Age < 80 years

Exclusion Criteria:

* Contraindication to sitagliptin or metformin or thiazolidinedione
* Pregnant or breast feeding women
* Type 1 diabetes, gestational diabetes, or secondary forms of diabetes
* Not appropriate for oral antidiabetic agent
* Medication which affect glycemic control
* Disease which affect efficacy and safety of drugs
* Any major illness (Liver disease, Renal failure, Heart disease, Cancer, etc)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change of HbA1c | 12 months
  Therapeutic efficacy of triple combination of metform, sitagliptin, and lobeglitazone compared with sulfonylurea and metformin in drug-naïve Korean type 2 diabetic patients

SECONDARY OUTCOMES:
beta-cell function | 12 months
  Changes of beta-cell function after one year treatment
Insulin resistance | 12 months
  Changes of Insulin resistance after one year treatment
Glucose homeostasis | 12 months
  Changes in fasting glucose concentration
Glucose metabolism | 12 months
  Area under the curve of glucose during OGTT
Glucose metabolism | 12 months
  Area under the curve of insulin during OGTT
Microalbuminuria | 12 months
  urine microalbumin to creatinine ratio
Lipid profile | 12 months
  Changes in TG/HDL/LDL-concentrations

OTHER OUTCOMES:
Hypoglycemia | 12 months
  Incidence of hypoglycemia during study period
Body weight | 12 months
  Changes of body weight after one year treatment
Body composition | 12 months
  Changes of body composition after one year treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea